| Protocol Title: |
|------------------------------------|
| Principal Investigator: |
| Site Principal Investigator: |
| Description of Subject Population: |

### About this consent form

Please read this form carefully. It tells you important information about a research study. A member of our research team will also talk to you about taking part in this research study. People who agree to take part in research studies are called "subjects." This term will be used throughout this consent form.

If you decide to take part in this research study, you must sign this form to show that you want to take part. We will give you a signed copy of this form to keep.

# **Key Information**

Taking part in this research study is up to you. You can decide not to take part. If you decide to take part now, you can change your mind and drop out later. Your decision won't change the medical care you get within [insert site name] now or in the future.

The following key information is to help you decide whether or not to take part in this research study. We have included more details about the research in the Detailed Information section that follows the key information.

# Why is this research study being done?

You are being asked to take part in this research study because you have immunoglobulin G4-related disease (IgG4-RD) that is currently active. The purpose of this study is to better understand the safety and side effects of an investigational drug called elotuzumab and to find what dose to use in people with IgG4-RD.

# How long will you take part in this research study?

This is Part 1 of a planned 2-part study. No one participates in both parts. Part 1 is testing the safety of two different dosing schedules of elotuzumab. This is a 1-year study for people with active IgG4-RD. Part 1A of the study enrolled 6 participants as planned to test a weekly schedule of a study drug called elotuzumab given by IV infusion each week for 4 weeks (total of

4 doses). An oral corticosteroid (Prednisone) taper was started at the time of the first dose that was finished in 10 weeks. A safety review was conducted when the 6<sup>th</sup> person finished his/her infusions and Prednisone taper. No safety concerns were identified and now we are moving to Part 1B. In this part 6 additional participants will be enrolled and given a different schedule of IV elotuzumab, which will be administered as an infusion every 2 months for a total of 6 doses. The Prednisone taper will be given the same way as in Part 1A. The purpose of the more spread- out doses is to continue to evaluate safety of the study drug while looking at its durability (long term effect) on IgG4-RD. During this time, we will ask you to visit the study site about once a month (16 visits).

## What will happen if you take part in this research study?

If you decide to join this research study, the following things will be done at various times in the study: physical exam, study drug infusions though an IV catheter, blood sample collection, urinalysis and urine pregnancy testing, possible CT (computed tomography) or MRI (magnetic resonance imaging) imaging, and have you fill out surveys about your health.

## Why might you choose to take part in this study?

We cannot promise any benefits to you from taking part in this research study. However, if you do receive elotuzumab, some of your IgG4-RD symptoms could possibly improve. Others with IgG4-RD may benefit in the future from what we learn in this study.

## Why might you choose NOT to take part in this study?

Taking part in this research study has some risks and requirements that you should consider carefully. This is a research study of an investigational drug that will be tested for the first time in patients with your disease. Side effects of elotuzumab reported in cancer patients include infusion reaction, infection, and liver problems. This study will use a less intensive treatment period than what is used to treat cancer. To try to reduce the risk of a reaction to elotuzumab, pre-medications will be given before each infusion, and you will be carefully monitored. As with all medications, there can be side effects. A detailed description of side effects can be found later in this consent form in the section called "What are the risks and possible discomforts from being in this research study?" Other things to consider are travel commitments for clinic visits. This study also involves at least 1 phone call visit where we will check in with you over the phone and/or computer after the first infusion to see how you are doing. If it is thought necessary for your health and well-being you may be asked to visit the study site for an unscheduled visit for a safety check.

# What other treatments or procedures are available for your condition?

You do not have to take part in this research study to be treated for IgG4-RD.

There is no cure for IgG4-RD. However, there are medications, such as glucocorticosteroids (prednisone) available to manage some symptoms of IgG4-RD. Alternative options that may be available to you include treatment with other medicines for IgG4-RD such as rituximab.

Talk with the study doctor if you have questions about any of these treatments or procedures.

# If you have questions or concerns about this research study, whom can you call?

You can call us with your questions or concerns. Our telephone numbers are listed below. Ask questions as often as you want.

| Dr. John Stone is the person in charge of | | | |
|---|---|---|---|
| M-F 9-5. You can also call Dr. | or Dr. | at ( | M F 9-5 |
| with questions about this research study. | You can also call p | age Dr. | or Dr. |
| at ( 24/7. | | | |
| If you have questions about the scheduling coordinator at | g of appointments | or study visits, call th | e study |
| If you want to speak with someone <b>not</b> di | rectly involved in | this research study, pl | ease contact |

You can talk to them about:

- Your rights as a research subject
- Your concerns about the research
- A complaint about the research
- Any pressure to take part in, or to continue in the research study

the Mass General Brigham IRB. You can call them at 8

### **Detailed Information**

A description of this clinical trial will be available on *http://www.ClinicalTrials.gov*, as required by U.S. Law. This website will not include information that can identify you. At most, the website will include a summary of the results. You can search this website at any time.

IgG4-RD is a chronic inflammatory and fibrotic condition that can affect virtually every organ system in the body. Some systems commonly affected are the pancreas, bile ducts, salivary and other glands and lymph nodes, peri-orbital area (around the eyes), lungs and kidneys. Over time, the inflammation becomes a more fibrotic "hardened, like scarring" condition that can lead to tissue damage and eventual organ failure if not treated.

Current treatment for IgG4-RD is primarily with corticosteroids (prednisone, methylprednisolone and others). While this approach is initially successful in most patients, the relapse rate is high when corticosteroid treatment is stopped. It is well-known that corticosteroids have side effects and long-term toxicities including glucose intolerance/diabetes, hypertension, weight gain, osteoporosis, increased risk of infection, glaucoma, cataracts and mood swings. More targeted treatments with other immunosuppressive drugs have been studied in small trials but no drug is approved by the U.S. Food and Drug Administration (FDA) for the treatment of IgG4-RD.

Elotuzumab targets the immune system, and specifically the B and T cells thought to be active in IgG4-RD. The drug targets SLAMF7, a protein found on cells of the immune system thought to be a key factor to the development of IgG4-RD. Elotuzumab is currently approved by the U.S. FDA for the treatment of a type of blood cancer called multiple myeloma. Elotuzumab has not been studied in IgG4-RD or any other autoimmune disease until now. For Ig4-RD the drug is experimental and can only be used in research studies.

This is Part 1 of a planned 2-part study. Part 1 is testing the safety of two different dosing schedules of Elotuzumab. This is a 1-year study for people with active IgG4-RD. Part 1A of the study enrolled 6 participants as planned to test a schedule of a study drug called elotuzumab given by IV infusion once weekly for 4 weeks (total of 4 doses). An oral corticosteroid (Prednisone) taper was started at the time of the first dose and was finished in 10 weeks. A safety review was conducted when the 6<sup>th</sup> person finished his/her infusions and Prednisone taper. No safety concerns were identified. We are moving to Part 1B. In this part 6 additional participants will be enrolled and given a different schedule of IV Elotuzumab, which will be administered as an infusion every 2 months for a total of 6 doses. The Prednisone taper will be given the same way as in Part 1A.

The purpose of the more spread- out doses is to continue to evaluate safety of the study drug while looking at its durability (long term effect) on IgG4-RD. You will be in the study for about 1- year from the time you join. During this time, we will ask you to visit the study site about once a month (16 visits). Some of these visits will be to administer the study drug. At all of the visits we will evaluate your overall health and IgG4-RD status.

If no safety concerns are seen, a larger Part 2 study is planned to look at elotuzumab effects in IgG4-RD.

The study is supported in part by a grant from the National Institute of Allergy and Infectious Diseases, of the National Institutes of Health (NIAID, NIH). Bristol-Myers Squibb Company (BMS) is the pharmaceutical manufacturer of elotuzumab providing the drug.

# Who will take part in this research?

About 6 participants will be entered in Part 1B of the study at one of approximately 3 centers in the U.S. with experience in treating IgG4-RD.

## What will happen in this research study?

During the study, you will participate in the following:

- Screening phase to see if you meet the requirements to participate.
- Treatment phase where you will receive the 12-month dosing schedule. We will also evaluate the safety of the study drug and your IgG4-RD with visits scheduled about once a month until the end of the study.

## **Background Medications and Vaccinations:**

These are drugs that will be given during the study in addition to the investigational drug.

### **Immunosuppressive Drugs:**

You will take oral prednisone at the beginning of the study that will be tapered off by 10 weeks after your first dose of elotuzumab. Depending on your disease status at the time you enter the study you may be started on up to 60 mg prednisone daily during the screening period. The dose will need to be decreased to 40 mg or 30 mg prednisone /day (depending on the dose you are taking if any) by the time you start the elotuzumab, which your study physician will manage with you. You should never abruptly stop or try to manage your prednisone taper on your own. If you have already been on prednisone 40 mg/day for at least two weeks during the screening period, then your prednisone dose will be 30 mg/day on the day of your first elotuzumab infusion.

The study will supply the daily oral prednisone beginning on the day of your first elotuzumab infusion through the end of the taper 10 weeks later.

If you are taking drugs other than corticosteroids (prednisone) to treat your IgG4-RD, you will be asked to taper off those medications during the screening period. It is possible that your IgG4-RD symptoms may worsen during this period. If screening procedures show that you fit all study criteria you will return to begin study treatment.

### **Prophylaxis for SARS-CoV-2 per CDC Guidelines:**

If you agree to participate you may receive medicines to help prevent SARS-CoV-2 if available and recommended by CDCat the time you enter the study.

Prophylaxis recommendations are subject to change over time depending on the state of the pandemic and prominent strain(s) of the virus. Your study doctor will inform you of the most up to date NIH/CDC recommendations.

(https://www.covid19treatmentguidelines.nih.gov/overview/prevention-of-sars-cov-2/)

#### **Vaccinations:**

Vaccination against the SARS-CoV-2 virus is required to participate in this study. Vaccination status must conform to CDC recommendations for immunocompromised individuals. Vaccination must have been completed at least 2 weeks prior to start of study therapy. These

recommendations are subject to change but are updated at:

https://www.cdc.gov/coronavirus/2019-ncov/vaccines/recommendations/immuno.html.

It is also recommended that you be up to date on receipt of other vaccinations to prevent infection before coming into the study. This includes the varicella zoster (Shingles) vaccine, the influenza (flu) vaccine, and the pneumonia vaccine.

If you have questions, your study doctor will discuss this with you.

### **Screening Phase**

Once you have signed the consent form, you will have a screening evaluation. A full medical history will be taken including the medications you take. This includes your routine cancer screening history. The screening evaluations are:

- Complete Physical Exam: including height, weight and vital signs-temperature, blood pressure, heart rate, and breathing rate.
- Routine Blood Tests: about 2 tablespoons of blood and a urine sample are collected to evaluate your disease status and overall health. This includes infectious disease testing for HIV, tuberculosis, and hepatitis. A pregnancy test is done for women able to become pregnant.
  - Research Blood Tests: an additional 2 tablespoons of blood are drawn for studies to look at your immune system and the effect of the study drug. We will collect a urine sample to test for your general health.
- Imaging Studies: A Computed Tomography (CT) scan is obtained to evaluate the organs affected by your IgG4-RD. This involves a series of detailed x-ray pictures while lying on a table.
  - o If you have had a recent CT scan, then Magnetic Resonance Imaging (MRI) may be substituted prior to treatment to limit your radiation exposure. MRI is a noninvasive test that uses a magnet to show detailed pictures of your organs. You lay on a table that moves into the cylinder-shaped tube where the pictures are taken. You are not exposed to x-rays for this. The MRI makes loud banging noises as it takes pictures. You are given earplugs or headphones and the technician can see, hear, and talk with you during the test.
  - Just before these procedures you may be given a substance called a contrast agent by injection into a vein. The contrast agent makes it easier to see different structures inside your body
- Optional Salivary Gland biopsy (MGH participants only\* Described later)

The screening visit takes about 2 hours plus the time for radiology imaging studies which may be done on a different day. Procedures may be scheduled over more than one visit within a 1-month period.

### (CT) Computed Tomography scan

Computerized tomography (CT) may be done. Just before these procedures, you may be given a substance called a contrast agent by injection into a vein. The contrast agent makes it easier to see different structures inside your body. Ultrasound may be done in subjects with abnormalities of the liver and/or pancreas.

### (MRI) Magnetic resonance imaging

MRI (magnetic resonance imaging) is a test that uses special equipment to take detailed pictures of body tissues and organs. During an MRI, you will lie very still, because any movement may make the pictures blurry, and the study doctor will not be able to interpret and understand the pictures. The MRI may also require a contrast agent injection to make it easier to see different structures inside your body.

### **Optional Submandibular gland (MGH only)**

An optional submandibular gland biopsy will be performed between screening and Baseline Day 0 and between Weeks 40 and 44 to assess the tissue response to study treatment. The subject will be instructed to stop aspirin or NSAID (medicines that are widely used to relieve pain, reduce inflammation, and bring down a high temperature) medication 3-7 days before the procedure. A local pain-killing medicine (anesthetic) may be injected, and a needle is inserted into the gland. A piece of tissue or cells are removed and placed on slides. An ice pack is then placed on the skin in the area of the biopsy to reduce swelling and bruising.

Dr. Ambrose Huang, from Interventional Radiology at MGH, will perform the submandibular gland biopsies.

| I agree to participation in optional submandibular gland biopsy. □ YES □ NO Initial | |
|---|---|
| After the results of the screening tests are available, the study doctor will determine if you qualify for this study. If you don't qualify, your study doctor will explain the other options the are available to manage your IgG4-RD. | ıat |

### **Treatment Phase**

You will be given a COVID-19 antigen self-test to take at home within 24 hours of each study drug infusion visit. This test is a nasal swab using a Q-Tip to swab the lining of both nostrils. Taking the test and getting the results takes about 15 minutes. You will be given clear instructions on how to perform the test and how to report the results.

### Baseline Visit (Visit 2)

If you qualify, you will return to the clinic to get your first IV dose of study drug. The study staff will discuss with you when the study treatment visits will occur.

Visit 2 will take about one hour. At this visit, we will:

- You will have your medical history and the list of medications that you take updated.
- You will be asked to report possible side effects.
- You will have vital signs taken including height and weight
- Physical Exam: a brief physical exam at each visit
- Draw a blood sample
  - O Safety Blood and Urine Tests: about 1½ teaspoons of blood will be drawn at each visit to look at your disease status and overall health
  - Research Blood Tests: an additional 2 tablespoons of blood are drawn for studies to look at your immune system and the effect of the study drug. Ask you for a urine sample for general health.
- Urine test for pregnancy, if you are a female who can become pregnant
- You will be asked to complete questionnaires and paper scale of disease activity

### Premedication

Before every dose all participants will receive pre-medications to help prevent an infusion reaction to the study drug while and just after it is given IV. These pre-medications are:

- an IV corticosteroid,
- famotidine (Pepcid® or equivalent) oral or IV,
- diphenhydramine (Benadryl® or equivalent) oral or IV,
- and an oral anti-fever medication (Tylenol®, acetaminophen).

## **Taking the Study Drug**

We have completed Part 1A of the study. In Part 1B, you will receive one elotuzumab infusion every 2 months for a total of 6 doses.

You are admitted to the infusion center on the mornings of each scheduled dose. After completion of the pre-infusion procedures (described below) you will have an IV catheter (thin, plastic tube) inserted in a vein in your arm or hand. Each dose of study drug is given over about 2 hours, and you are closely monitored for safety during and after the infusion. You should plan to be in the infusion center for approximately 4-6 hours on each of the infusion days.

### Prednisone Taper

On the first infusion day, you will begin taking prednisone every day for a 10- week taper. You will start at 40 mg prednisone/day unless you have already been taking this dose for at least 2 weeks prior. If so, you may begin the taper at prednisone 30 mg/day. This will be provided by the study in bottles with clear instructions for how to taper the dose. You are asked to bring your

bottles back to each study visit. Each dose is in a different bottle with a different color capsule. You will be given multiple bottles with clear instructions on when to start and stop each bottle. There will be extra capsules in each bottle to return at your next scheduled study visit. Site study staff will explain how to take the prednisone in a decreasing dose over the next 10 weeks until you have finished the taper and are taking no more. Please do not take your morning dose on the day of any study visit, as you will take that day's dose from the new bottle given to you.

#### **Part 1B Treatment Phase**

The study visits are scheduled about monthly, with the study drug administered every 2 months for 6 doses. You will visit the study site for safety checks where you don't receive the study drug in between. A phone/virtual visit will be conducted about 7 days after your 1<sup>st</sup> infusion to see how you are doing. If thought necessary for your safety/well-being you may be asked to come in for an unscheduled visit. For the 12-month treatment schedule the infusions happen at Week 0 (1<sup>st</sup> dosing visit), and again at Weeks 8, 16, 24, 32, & 40)

The final study visits for safety and status of your IgG4-RD happen at Weeks 44 and 48 (about one year after starting).

### Each In person Visit

At each visit during this part of the study, the following will happen:

- We will review your medications
- You will be asked to report possible side effects.
- You will have vital signs taken including height and weight
- You may have a physical examination by the study doctor
- Safety Blood and Urine Tests: About 1½ teaspoons will be drawn for this health check at the safety visits and within 48-72 hours of each study drug infusion visit.

#### Most Visits

At most visits, we will also obtain/perform:

- A brief physical exam at each visit except for the Week 24 and 48 visits, when you have a complete physical exam.
- You will be given a COVID-19 antigen self-test to take at home within 24 hours of each study drug infusion visit. This test is a nasal swab using a Q-Tip to swab the lining of both nostrils. Taking the test and getting the results takes about 15 minutes. You will be given clear instructions on how to perform the test and how to report the results. (Wks. 8, 16, 24, 32, & 40)
- Urine test for pregnancy if you are a female who can become pregnant (Wks. 8, 16, 24, 32, & 40)
- Draw a blood research blood test: an additional 2 tablespoons of blood are drawn for studies to look at your immune system and the effect of the study drug (approximately every 2 months).

- Ask you for a urine sample for general health ((3 times during the study)
- Premedication and study drug infusion (Wks. 8, 16, 24, 32, & 40)
- You will be asked to complete questionnaires and paper scale of disease activity

#### Some Visits

At some visits, we will:

- Complete physical exam (Wks. 24 & 48)
- Obtain imaging Studies: CT scan or MRI is repeated to evaluate the organs affected by your IgG4-RD at the Week 48visit. The follow-up visits should take about one hour, except for the Week 48 visit which can take 3-4 hours, depending on time needed for CT/MRI
- Review prednisone taper (Wks. 1(by phone), 4, 8, &12) Extra or unplanned visits

You may be asked to return to the study site in-between the visits described above if your study doctor thinks it important for your safety.

### **After You Complete the Study**

After you complete the study, we will refer you back to your own doctor for your ongoing medical care.

### **Stopping the Study Early**

You may have study drug discontinued without your consent at any time. Reasons why this could happen include, but are not limited to, the following:

- Your study doctor decides that it is best for you not to continue.
- You are unable to complete study tests.
- The study is stopped by the Institution, the Sponsor(s), or other health authorities.
- You become pregnant or plan to get pregnant during this study.
- You have severe side effects from elotuzumab.
- You need medications that are not allowed for this study.
- Your disease gets worse in the kidney or in other organs.

If study drug is discontinued early, we would like for you to continue all follow-up visits through one year. Otherwise, we would like to see you for a study discontinuation visit which will include all assessments listed for the Week 48 visit.

# How may we use and share your samples and health information for other research?

#### Health Information

Your medical and research records will be confidential to the extent permitted by law. Every effort is made to keep your identity private. However, we cannot guarantee complete confidentiality.

You will be identified by a study code, not your name. Personal information from your records will not be released without your written permission. You will not be identified in any publication or in the sharing of your data about this study. After the study is completed, this study data may be placed in a central storage location. These data will not include your name or other information that can identify you. The purpose is to make study data available to other researchers. Information from this study may be put into databases along with information from other studies. There are different kinds of databases; some are publicly accessible, and some are restricted. Only researchers who apply and are approved can access restricted databases. Traditionally used identifying information about you (such as name, address, medical record #, etc.) will NOT be included or shared with others.

In an NIH funded study, you are further protected through a policy that prevents the study doctor from releasing any sensitive information about you that may identify you. This would not prevent you or a family member from voluntarily releasing information about this research. Organizations that may look at and/or copy your medical records for research, quality assurance, and data analysis include:

- The National Institute of Allergy and Infectious Diseases (NIAID, NIH), sponsor of this research;
- o NIAID representatives, agents, employees, contractors, grantees and other persons assisting in the conduct, monitoring, or analysis of this study;
- o Representatives of Bristol-Myers Squibb, Co., the pharmaceutical partner providing the study drug
- o The U.S. Food and Drug Administration (FDA);
- Other state and local health and/or regulatory authorities.

These organizations and agencies may also ask permission to look at your medical records from other doctors, hospitals, or other healthcare providers.

After the study is completed, the data are placed in a central storage location, or public database. This includes all the information learned from this study and not just information about you. The reason is to share data with other researchers. All data is coded and will not be linked with your name or other identifying information such as social security number or birthday.

#### OPTIONAL STORAGE OF LEFTOVER BLOOD SAMPLES FOR FUTURE USE

We would like to ask your permission to store any left-over blood from the samples collected to be used in the future to study the immune system, IgG4-RD, and other diseases. Since we do not yet know the exact questions that will be studied, we cannot tell you exactly what tests will be

done on your samples. As a research participant in this study, you have the option of allowing any leftover blood samples to be stored for future tests. Samples will be stored at the Ragon Institute of MGH, MIT and Harvard, and at Emory University. We plan to store your samples for an unknown length of time.

We may want to share your samples with researchers at other institutions. Your samples will be coded with a number so that your name cannot be identified. Only the investigators of this study will have the code that links you to your specimens. Reports about research done with your samples will not be put in your medical record and will be kept confidential, to the best of our ability and within state and federal law. Information that does not become part of your medical record will be identified by a code, and personal information from your records will not be released without your written permission. You will not be identified in any publication about this study. Reports on these stored samples will not be given to you or your physician(s). Your blood samples will not be sold or used directly to produce commercial products.

You can change your mind at any time and ask to have your samples destroyed, and we ask that you notify your study physician in writing if you choose to do so. If your sample(s) have not been used for future tests, they will be destroyed when your request is received. If your sample(s) have already been used prior to this request, then the information will be used in the overall study analysis.

Benefits: There are no direct benefits to you from the collection and storage of these samples. The benefit of research on stored samples for society is the information that can be learned about the immune system and IgG4RD. You will not receive any financial gain from studies done using your stored samples.

Risks: There may be unknown risks associated with the storage and analysis of your blood samples or the information resulting from the analysis of your samples. Every effort will be made to maintain your confidentiality.

Making a Decision: Please consider the storage of leftover blood samples for future use as described above and answer the question below. No matter what you decide, it will not affect your care or participation in this study. The choice is up to you.

| Please indicate | your | response | below: |
|-----------------|------|----------|--------|
|-----------------|------|----------|--------|

| sharing of in planned. | _ | ing of my samples (blood, tissue (MGH biopsies)) and a those future analyses for genetic tests not currently |
|---|---|---|
| I agree to the | e storage, future use and shari | ing of my samples (blood, tissue) and sharing of ure analyses for other tests not currently planned. |
| □ YES □ N | O Initial | |
| <u>OPTIONAI</u> | L FUTURE CONTACT | |
| contact you is as a follow-u | in the future related to your he<br>up to this study or we may con | your study doctor would like to ask your permission to ealth and participation in this study. We may contact you tact you to invite you to take part in future studies related below whether you would allow future contact by us. |
| Please initia | l/date your responses to the j | following questions below: |
| I agree to pe RD. | rmit my study doctor to conta | act me regarding future research studies related to IgG-4 |
| □ YES<br>□ No | Initial | Date:/_/ Date:// |
| - | rmit a study doctor to contact s study after my participation | t me in the future as a follow-up to my health status has ended. |
| □ YES<br>□ No | Initial<br>Initial | Date:// Date:// |
| | t the results of this research | |

Caparally, we will not give you or your doctor information about

• Generally, we will not give you or your doctor information about the results of your individual participation in the research study. The research we are doing is only a stepping-stone in understanding IgG4. Most of the findings that come from studying your samples or

- information will not be relevant to your personal health. However, in the future, this may change.
- It is important to remember that research results are not always meaningful and are not the same as clinical tests. While you should not expect to get any information about the results of your participation in this research, if something about you is learned that would be important for you to know for your safety or well-being, we will attempt to contact you to let you know. In some situations, follow-up testing might be needed. in a certified clinical lab. You and your medical insurer will may be responsible for the costs of these follow-up tests and any follow-up care, including deductibles and co-payments.

# What are the risks and possible discomforts from being in this research study?

**Elotuzumab Risks** 

### **Infusion Reaction**

The information on risks and side effects with elotuzumab from the drug manufacturer, Bristol-Myers Squibb Company, comes from the cancer studies in multiple myeloma. There have been reports of infusion reactions in up to 10% of patients in the large trials, with 70% happening during the first dose. The most common symptoms of an infusion reaction included fever, chills, and low blood pressure. Other symptoms may include the following: rash, chest pain, trouble breathing, swelling of the throat/tongue (extremely rare allergic reaction), dizziness, light-headedness. Most of the reactions were mild or moderate, resulting in temporary stopping of the infusion to treat the reaction. 1% were severe resulting in permanent discontinuation of the drug. While there have been no reports of life-threatening reactions, there is the potential for serious, life-threatening reactions including anaphylaxis (severe allergic reaction).

Infusion reactions can happen during the elotuzumab infusion or within 24 hours after. Before every infusion, you will receive pre-medications to help lower your chances of having an infusion reaction. These include:

- glucocorticoids that you will receive intravenously,
- diphenhydramine (Benadryl®/equivalent) intravenously or orally,
- famotidine (Pepcid® or equivalent) intravenously or orally, and
- acetaminophen (Tylenol®/equivalent) orally.

You will be monitored closely by the research team during and after the infusions who are trained and equipped to quickly manage a reaction. If needed the drug will be temporarily stopped and/or the rate slowed down.

#### Other Frequently reported Adverse Events

- fatigue
- numbness

- weakness
- tingling
- burning pain in your arms or legs
- diarrhea
- sore throat or runny nose
- fever
- upper respiratory tract infection
- constipation
- decreased appetite
- cough
- pneumonia

### Infection

Infections have been reported in the cancer studies occurring in most patients. Some of these infections were severe or life-threatening resulting in hospitalization. Fatal infections were rare. The most common serious infections were pneumonia and respiratory tract infections. Other unusual infections reported included fungal infections (10%), and herpes zoster (17%). Make sure you contact your study doctor and seek medical care right away if you have any signs and symptoms of an infection, including fever, flu-like symptoms, sore throat, cough, shortness of breath, burning with urination, a painful skin rash, or other.

Before coming into the study you are encouraged to be up-to-date on recommended vaccinations to prevent infection, including the varicella zoster (Shingles) vaccine. Your study doctor will discuss this with you if you have questions.

### Liver Damage (Hepatotoxicity)

One of the large cancer studies reported increases in liver function blood tests in small numbers of people. Some resulted in discontinuation of treatment, but most did not.

In this study you will be monitored closely with frequent blood tests to check your liver. The elotuzumab may be discontinued if needed for your safety. Inform your study doctor and seek medical care right away if you have signs and symptoms of liver problems including tiredness, weakness, loss of appetite, yellowing of your eyes or skin, color changes in your stools, confusion, or swelling of the stomach area.

#### Cancer (Malignancy)

Studies with the drug have been in cancer (multiple myeloma). There are no reports showing safety concerns of development of new cancers in these trials. As a precaution, this study will not enroll people who had cancer in the past 5 years (except for successful treatment

(excision) of cervical and non-myeloma skin cancer). If over the age of 50 (and earlier if you have risk factors) you should have age-appropriate cancer screenings prior to participating and throughout the study. Inform your study doctor and health care provider right away for any warning signs of cancer. More information may be found on the American Cancer Society website: http://www.cancer.org/healthy/find-cancer-early/cancer-screening-guidelines.html

There may be unanticipated risks which we are not yet aware of. You will be informed of any new risk information as we learn of it.

There may be other unknown risks from taking elotuzumab that we do not know about yet.

## Corticosteroid/prednisone Risks

Common side effects of corticosteroids used for a daily tapering dose as we will prescribe include glucose intolerance/diabetes, hypertension, osteoporosis (thinning of bones), increased risk of infection, glaucoma, cataracts, weight gain, moon face, acne, thin skin, mood swings, and irritability. The risk of the more permanent effects increases with chronic, longer-term use.

### Pre- Medication Risks

Risks of the pre-medications administered to decrease the risk of study drug infusion reaction are listed in the table below. The corticosteroid side effects described above related to daily dosing do not all apply to the single doses given as pre-medication. Those more short-term effects are described below.

- Corticosteroids/glucocorticoids: Mood swings, hot flashes, insomnia
- famotidine (Pepcid® or equivalent): Headache, constipation, nausea, vomiting, diarrhea
- acetaminophen (Tylenol/equivalent): Rash, nausea, headache; very rarely: hypersensitivity (allergic reaction), serious skin reactions, kidney/liver damage with high doses or drug/alcohol interactions
- diphenhydramine (Benadryl/equivalent): Somnolence (drowsiness), difficulty concentrating, dry mouth, difficulty urinating, constipation

### **Study Procedure Risks**

### **Blood Drawing Risks**

Possible side effects from having blood drawn include dizziness, redness and swelling of the vein, pain, bruising, or bleeding from the site of the needle puncture. There is also a chance of infection.

## **Blood collection during study:**

The following table shows the amount of blood that will be taken from you at each visit

| Visits | Amount of blood withdrawn |
|-------------------------------|-------------------------------------------|
| Screening | Approximately 27 mL (about 2 tablespoons) |
| Baseline | Approximately 78 mL (about 5 tablespoons) |
| Weeks 4, 12, 20, 28, 36, 44 | Approximately 7 mL (about 1½ teaspoons) |
| Weeks 8, 16, 24, 32, 40, & 48 | Approximately 57 mL (about 4 tablespoons) |

#### IV Catheter Risks

The risks for this procedure are rare and often mild. They include minor discomfort, bleeding, and bruising at the needle site. These symptoms often get better without medical help. You may also have some restriction of movement during the infusion time. Infection (indicated by redness, warmth, pain, swelling, and foul-smelling discharge) at the needle site can rarely occur.

### Optional Submandibular Gland Biopsy

Risks from this procedure may include:

- Allergic reaction to the anesthetic
- Bleeding
- Infection
- Injury to the facial or trigeminal nerve (rare)
- Numbness of the lip

### **Radiation Risks**

CT (Computerized Tomography) Scan: As a result of your participation in this study you may be exposed to radiation from up to 2 CT scans. If you take part in this research protocol, you may undergo CT scans during screening involving ionizing radiation. These would not be needed for clinical care if you were not in the research study. The type and body parts included in the imaging studies will depend on your diagnosis. In general, exposure to ionizing radiation may have health risks. In clinical imaging studies the benefits to individual normally overweigh risks. In research studies the benefits are normally to future groups or population and may not be to the individual.

You will be exposed to a maximum of approximately 24 millisieverts (mSv) for this research. A mSv is a unit of radiation dose. This amount of radiation is about the same as you would normally get in about 8 years from natural background sources from the earth and the sky.

The radiation doses used in this study could cause a small increase in the risk of developing cancer later in life. We always try to use the smallest possible radiation dose needed to get the imaging information we need. If you are pregnant or breastfeeding, you will not be able to participate in this research study.

Since the effects of radiation can add up over time, it is important that you tell the study doctor about your past clinical imaging and research-related radiation exposure. If you have taken part in other research studies in the past 12 months that have involved radiation exposure, please tell us. If it appears that your earlier radiation exposure is more than our current guidelines, it is possible that you will not be allowed to participate in this study. Please initial next to your choice below:

| I <u>have</u> participated in other research studies (not including this study) involving radiation exposure within the last 12 months. |
|---|
| I have not participated in other research studies (not including this study) involving radiation exposure within the last 12 months. |

#### **CT Contrast Risks:**

It is possible that you may receive contrast material (dye like iodine) intravenously or barium to swallow for the CT scans. Contrast material may rarely cause an allergic reaction, or very rarely serious reaction (anaphylaxis). Let the study doctor know if you are allergic to shellfish or iodine or have had a reaction to contrast dye in the past. Contrast material can harm to the kidneys, particularly in people with kidney disease. If you have kidney disease related to your IgG4-RD or other cause, then use of contrast material may not be an option.

Risk of MRI Scans: MRIs use powerful magnets to make images. There are no known radiation risks associated with MRI. However, persons with metal implants, such as surgical clips, or pacemakers should not have an MRI. All credit cards and other items with magnetic strips should also be kept out of the MRI room. People who feel uncomfortable in confined spaces (claustrophobia) may feel uncomfortable in the narrow tube. The MRI makes loud banging noises as it takes images. Earplugs can be used to reduce the noises. The MRI can be stopped at any time at your request. If you are or suspect you are pregnant, you should not participate in this study. The MRI has the potential, during normal routine use, to cause localized warming of your skin and the underlying tissues. You should immediately inform us if you experience discomfort due to warming and the procedure will be stopped.

Some people experience dizziness or rarely nausea when going into an MRI scanner and these sensations may be more common in scans with higher magnetic fields. In most cases, these symptoms only last a short time. However, some people may experience them throughout the scan and/or continue to experience them for a short period of time after; generally, less than half an hour. No case of permanent problems is known.

### Gadolinium contrast Risks

No all subjects will receive gadolinium in this study. A few patients will report a cold feeling in the arm during the injection, which is of no significance. An even smaller number (between about 1 and 4 in 100) will notice mild nausea or headache. Vomiting can occur, but this is rare (less than 1 in 100 injections). Even less often, in approximately 1 in 1000 patients, an itchy skin rash might appear a few minutes after the injection. This appears to be due to a mild allergy. It usually settles down by itself within an hour or so, but rarely it might be a warning sign of a more serious allergic reaction developing.

Severe allergic (anaphylactic) reactions to gadolinium are rare. These severe reactions, which might involve difficulty breathing and swelling of the lips and mouth, occur in approximately 1 in every 10,000 people who have gadolinium. These severe reactions generally respond very well to standard emergency drug treatment, like that given for other severe allergic reactions. These are usually medications that will be given through the tube that was placed in your arm before or during the MRI scan.

#### **Vaccine Risks**

Both elotuzumab and corticosteroids blunt (decrease) your immune system's response which may decrease the amount of protection you receive from vaccines. For this reason, certain vaccines, including booster with the COVID-19 vaccine, must occur at least 2 weeks before receiving the first dose of study drug. This study drug may also increase your risk of infection after receiving a live vaccine (for example: mumps, measles, and rubella). You should not receive any live vaccinations for at least 30 days before you enter the study and for at least 3 months after your last dose of study drug.

We advise you to be up to date with all recommended vaccines at least 2 weeks before enrolling in this study.

## **Incidental Findings**

If during the study testing, unexpected (non-study-related) information is learned that would be important for you to know for your well-being, you will be informed. This includes findings from the radiology (CT or MRI) tests. Counseling will be provided on next steps to take. The study will not cover costs for related follow-up outside of the study.

### Information related to COVID-19

- Immunization with one of the FDA authorized or licensed SARS-CoV-2 vaccines is required for study entry. Vaccination series must have been completed at least 2 weeks prior to start of study therapy.
- Both elotuzumab and corticosteroids suppress your immune system and may increase your susceptibility to getting a COVID-19 infection. Also, infection could be more severe as a result of receiving these drugs. This is true with any infection when taking drugs that

- suppress the immune system. These drugs may also interfere with the amount of protection you receive from a COVID-19 vaccination.
- The COVID-19 public health emergency changed the study. Enrollment in the study was closed temporarily while safety measures were added to the protocol. Visits were conducted remotely or virtually in some cases. Changes were made to how the study was conducted. Though the pandemic is considered over, safety measures related to COVID-19 remain in place.
- Measures to protect yourself and others from COVID-19 infection are outlined on the
  Centers for Disease Control website at the following link:
  https://www.cdc.gov/coronavirus/2019-ncov/prevent-getting-sick/prevention.html. To
  decrease your risk of infection with SARS-CoV-2, we strongly recommend that you
  follow these recommendations, which include wearing a mask, practicing social
  distancing, and frequent handwashing/use of hand sanitizer.

If you develop COVID-19 infection during your participation in the study, the infusions of elotuzumab will be suspended until you have recovered from the infection.

### Risks to an Embryo or Fetus, or to a Breastfeeding Infant

The risks to a developing fetus or breast-feeding infant are unknown with this drug. You cannot participate in this study if you are pregnant, breastfeeding or planning a pregnancy while in the study.

Female participants of childbearing potential and male participants with a partner of childbearing potential must agree to use a highly effective method of contraception throughout the study, for 6 months after the last infusion of elotuzumab. Highly effective methods are defined as those, alone or in combination, with a low failure rate (i.e. less than 1 percent pregnancy per year) when used consistently and correctly. Options include implant or intrauterine device (IUD), other hormonal method (injectable, oral, transdermal) with barrier method, or double barrier method. If you leave the study early, you must use contraceptive methods for at least 6 months after your last dose of study drug. If you are a woman able to become pregnant, we will perform pregnancy testing throughout the study. You will be asked about your reproductive potential and contraceptive use at each visit.

If you should become pregnant while in this study, or if you think your partner is pregnant (male participant), you must contact a study doctor right away. If you are female and still receiving the study drug, the doctor will stop it and you will continue to be followed until the baby is born or the pregnancy is ended.

# What are the possible benefits from being in this research study?

There are no direct benefits to you to be in this study. What is learned from the study may benefit society and help others with IgG4-RD in the future.

## What other treatments or procedures are available for your condition?

You do not have to take part in this research study to be treated for IgG4-RD. There is currently no cure for IgG4-RD. However, there are medications, such as corticosteroids/glucocorticoids (prednisone) available to manage some symptoms of IgG4-RD. Alternative options that may be available to you include treatment with other medicines such as rituximab.

Talk with your study doctor if you have questions about any of these treatments.

You will be informed of any new findings from this or other research that may affect your willingness to continue in this study.

If, during the study testing, unexpected (not study-related) information is learned that would be important for you to know for your well-being, you will be informed of that information. Counseling will be provided as to next steps. The study will not cover costs for related follow-up.

# Can you still get medical care within [insert site name] if you don't take part in this research study, or if you stop taking part?

Yes. Your decision won't change the medical care you get within [insert site name] now or in the future. There will be no penalty, and you won't lose any benefits you receive now or have a right to receive.

We will tell you if we learn new information that could make you change your mind about taking part in this research study.

# What should you do if you want to stop taking part in the study?

If you take part in this research study, and want to drop out, you should tell us. We will make sure that you stop the study safely. We will also talk to you about follow-up care, if needed.

Also, it is possible that we will have to ask you to drop out of the study before you finish it. If this happens, we will tell you why. We will also help arrange other care for you, if needed.

## Will you be paid to take part in this research study?

For part 1, you will be paid \$1,500.00 if you complete the study. If you do not complete the study, we will pay you \$125 for each infusion visit and \$75 for non-infusion visits you complete.

| Visit | Stipend |
|--------------------------|----------|
| Infusion visits (6) | \$750.00 |
| Non-Infusion visits (10) | 750.00 |

We may use your samples and information to develop a new product or medical test to be sold. The Sponsor, hospital, and researchers may benefit if this happens. There are no plans to pay you if your samples or information are used for this purpose.

We may be using an approved, outside vendor (Forte Research to make these payments to you via a reloadable credit card-based system, called Forte Payments. This secure system is like a gift card or credit card.

If you are paid by this system, you will be given a Forte Payments Visa card when you enroll in the study. Once the card is activated, the study team will add a payment after each paid visit you complete. The payment should be available to you within a day. You may use the card anywhere Visa cards are accepted, such as at a grocery store.

All reasonable expenses related to travel to and from the study site including lodging, meals, and transportation will be reimbursed. Participating patients and/or families will need to provide receipts for travel reimbursement.

#### Part 1 B: All visits outlined in consent form

- Up to the government's per diem lodging rate for your area (see http://www.gsa.gov/portal/category/100120 for details)
  - A second day/night may be charged for Screening, Day 0, weeks 4, 8, 16, 24, 32, and 40Up to the government's per diem meals rate for your area (see http://www.gsa.gov/portal/category/100120 for details)
    - A second day/night may be charged for Screening, Day 0, weeks 4, 8, 16, 24, 32, and 40Up to \$50/visit for transportation for subjects who live 121-300 miles away → \$450 / subject
    - Up to \$600/visit for airfare for subjects who live more than 300 miles away  $\rightarrow$  \$5,400 / subject

We will need to collect your Social Security number in order to make these payments, and it will be shared securely with the company that runs the card-based system. Payments like this are considered taxable income. If you receive more than \$600, the payment will be reported to the IRS as income by the hospital. If you provide a receipt for something like travel expenses and we can cover that, that is not considered taxable income. Reimbursement of expenses will not be made using the Forte Payments card.

## What will you have to pay for if you take part in this research study?

Costs related to usual clinical care of your IgG4-RD or other medical problems will be billed to you and/or your insurance provider(s). The study drug, elotuzumab, is being provided by the manufacturer, Bristol-Myers Squibb, Co. The study is providing the pre-medications for the infusions and steroid tablets for the prednisone taper. Other clinical and professional services including diagnostic and laboratory tests that are a part of this study and not part of your regular care will be covered by the study.

# What happens if you are injured as a result of taking part in this research study?

We will offer you the care needed to treat any injury that directly results from taking part in this research study. We reserve the right to bill your insurance company or other third parties, if appropriate, for the care you get for the injury. We will try to have these costs paid for, but you may be responsible for some of them. For example, if the care is billed to your insurer, you will be responsible for payment of any deductibles and co-payments required by your insurer.

Injuries sometimes happen in research even when no one is at fault. There are no plans to pay you or give you other compensation for an injury, should one occur. However, you are not giving up any of your legal rights by signing this form.

If you think you have been injured or have experienced a medical problem as a result of taking part in this research study, tell the person in charge of this study as soon as possible. The researcher's name and phone number are listed in the beginning of this consent form.

## If you take part in this research study, how will we protect your privacy?

Federal law requires Mass General Brigham to protect the privacy of health information and related information that identifies you. We refer to this information as "identifiable information."

#### In this study, we may collect identifiable information about you from:

• Past, present, and future medical records

 Research procedures, including research office visits, tests, interviews, and questionnaires

### Who may see, use, and share your identifiable information and why:

- Mass General Brigham researchers and staff involved in this study
- The sponsor(s) of the study, and people or groups it hires to help perform this research or to audit the research
- Other researchers and medical centers that are part of this study
- The Mass General Brigham ethics board or an ethics board outside Mass General Brigham that oversees the research
- A group that oversees the data (study information) and safety of this study
- Non-research staff within Mass General Brigham who need identifiable information to do their jobs, such as for treatment, payment (billing), or hospital operations (such as assessing the quality of care or research)
- People or groups that we hire to do certain work for us, such as data storage companies, accreditors, insurers, and lawyers
- Federal agencies (such as the U.S. Department of Health and Human Services (DHHS) and agencies within DHHS like the Food and Drug Administration, the National Institutes of Health, and the Office for Human Research Protections), state agencies, and foreign government bodies that oversee, evaluate, and audit research, which may include inspection of your records
- Public health and safety authorities, if we learn information that could mean harm to you
  or others (such as to make required reports about communicable diseases or about child
  or elder abuse)
- Other researchers within or outside Mass General Brigham, for use in other research as allowed by law.

### **Certificate of Confidentiality**

A federal Certificate of Confidentiality (Certificate) has been issued for this research to add special protection for information and specimens that may identify you. With a Certificate, unless you give permission (such as in this form) and except as described above, the researchers are not allowed to share your identifiable information or identifiable specimens, including for a court order or subpoena.

Certain information from the research will be put into your medical record and will not be covered by the Certificate. This includes records of medical tests or procedures done at the hospitals and clinics, and information that treating health care providers may need to care for you. Please ask your study doctor if you have any questions about what information will be included in your medical record. Other researchers receiving your identifiable information or

specimens are expected to comply with the privacy protections of the Certificate. The Certificate does not stop you from voluntarily releasing information about yourself or your participation in this study.

Even with these measures to protect your privacy, once your identifiable information is shared outside Mass General Brigham, we cannot control all the ways that others use or share it and cannot promise that it will remain completely private.

Because research is an ongoing process, we cannot give you an exact date when we will either destroy or stop using or sharing your identifiable information. Your permission to use and share your identifiable information does not expire.

The results of this research may be published in a medical book or journal or used to teach others. However, your name or other identifiable information **will not** be used for these purposes without your specific permission.

### **Your Privacy Rights**

You have the right **not** to sign this form that allows us to use and share your identifiable information for research; however, if you don't sign it, you can't take part in this research study.

You have the right to withdraw your permission for us to use or share your identifiable information for this research study. If you want to withdraw your permission, you must notify the person in charge of this research study in writing. Once permission is withdrawn, you cannot continue to take part in the study.

If you withdraw your permission, we will not be able to take back information that has already been used or shared with others, and such information may continue to be used for certain purposes, such as to comply with the law or maintain the reliability of the study.

You have the right to see and get a copy of your identifiable information that is used or shared for treatment or for payment. To ask for this information, please contact the person in charge of this research study. You may only get such information after the research is finished.

## **Informed Consent and Authorization**

## **Statement of Person Giving Informed Consent and Authorization**

- I have read this consent form.
- This research study has been explained to me, including risks and possible benefits (if any), other possible treatments or procedures, and other important things about the study.
- I have had the opportunity to ask questions.
- I understand the information given to me.

## **Signature of Subject:**

| Subject | Date | Time |
|---|---|---|
| Signature of Study Doctor or Person | Obtaining Cons | ent: |
| Statement of Study Doctor or Person Obtain | ning Consent | |
| Statement of Study Doctor or Person Obtain I have explained the research to the study | S | |
| <ul> <li>I have explained the research to the students.</li> <li>I have answered all questions about this</li> </ul> | dy subject. | the best of my ability. |